CLINICAL TRIAL: NCT03442127
Title: Facilitating Oncology Patient-Clinician Communication Via E-health Innovations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0432-17-EP
Record Dates: First submitted 2018-02-02; First posted 2018-02-22 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Group (Other): Program users
  Interventions: Behavioral: CaringGuidance™ After Breast Cancer Diagnosis

INTERVENTIONS:
Behavioral: CaringGuidance™ After Breast Cancer Diagnosis — Web-based, psychoeducational, self-management tool

SUMMARY:
The Internet-based program CaringGuidance™ After Breast Cancer Diagnosis and its new electronic Summary Report (CGSR) tool are hypothesized to empower patients to raise their emotional and social concerns during oncology consultations and assist medical oncology clinicians in identifying patient needs. This study will assess satisfaction and feasibility of clinical use of the new patient guided, Internet-based CGSR to support patient-clinician communication in the outpatient breast oncology clinic. Participants will have access to the CaringGuidance™ program for home use on computer or mobile device. Following this, paricipants will meet with an investigator prior to a medical oncology appointment and create a CGSR on an iPad while they talk through the process. These assessments will help characterize the emotional state at the time of working with the program and the CGSR. Participants will take the CGSR into their oncology appointment, record the appointment if she and the physician have consented to this, and use the CGSR as much or as little as desired. Data will be analyzed primarily qualitatively to determine participant's appraisal of the functionality, content satisfaction and usability of the CGSR and communication patterns, topics discussed during the appointment and patient/clinician satisfaction with communication during the appointment when the CGSR was available for use.

DETAILED DESCRIPTION:
The Internet-based program CaringGuidance™ After Breast Cancer Diagnosis and its new electronic Summary Report (CGSR) tool are hypothesized to empower patients to raise their emotional and social concerns during oncology consultations and assist medical oncology clinicians in identifying patient needs. The purpose of this study is to assess satisfaction and feasibility of clinical use of the new patient guided, Internet-based CGSR to support patient-clinician communication in the outpatient breast oncology clinic. The study will enroll 30 women who are being treated for breast cancer. They will all have access to the CaringGuidance™ program for at home use on computer or mobile device for approximately one month (or up to 6 months depending on when they return to their primary medical oncologist for evaluation). Following this, these women will meet with the researcher or research assistant prior to a medical oncology appointment and create a CGSR on an iPad while they talk through the process with the researcher. Women will complete demographic data and assessment of coping prior to receiving access to the program and at this appointment. These assessments will help characterize the emotional state at the time of working with the program and the CGSR, these measures are not to assess the efficacy of the program. Clinicians will complete a brief, one-time demographics survey prior to enrollment of patients to the study. Women will take the CGSR into their oncology appointment, record the appointment if she and the physician have consented to this, and use the CGSR as much or as little as desired. Clinicians will complete a brief satisfaction survey following the appointment and patients will debrief (recorded) about whether they used the CGSR and their impressions following the appointment. Data will be analyzed primarily qualitatively to determine women's appraisal of the functionality, content satisfaction and usability of the CGSR and the communication patterns, topics discussed during the appointment and patient/clinician satisfaction with communication during the appointment when the CGSR was available for use. Data will be used for future modification of the CGSR to assure that it meets patients' needs prior to initiating a larger scale trial.

ELIGIBILITY:
Inclusion Criteria:

* first, stage I - IV breast cancer
* have had at least 1 appointment with a medical oncologist with additional -appointments planned at University of Nebraska Medical Center/Nebraska Medicine clinics,
* able to read and speak English,
* have regular access to Internet and computer,
* have email

Exclusion Criteria:

* Male,
* mentally or physically unable to consent or use the CaringGuidance program (e.g. hospitalized in the past year with a substance abuse or mental health condition)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction with the Content of the CaringGuidance Summary Report Form | 1 minute
  qualitative description from the patient regarding their satisfaction with the content of the CaringGuidance Summary Report
Functionality of the CaringGuidance Summary Report Form | 10 minutes
  qualitative description of the functioning of the CaringGuidance Summary Report
Usability of the CaringGuidance Summary Report From | 20 minutes
  quantitative measure of usability of the form by the System Usability Scale a 10 item scale (strongly disagree to strongly agree) developed by John Brookes 1986 at Digital Equipment Corporation and used in multiple studies.The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking.
  Based on research, a System Usability Scale score above a 68 would be considered above average and anything below 68 is below average, however the best way to interpret your results involves "normalizing" the scores to produce a percentile ranking.

SECONDARY OUTCOMES:
Patient-clinician communication using CaringGuidance Summary Report Form | during clinical encounter, approximately 20 minutes
  qualitative description of psychosocial topics discussed

CONTACTS AND LOCATIONS:
Overall Officials: Robin M Lally, PhD, RN, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Oncology Clinics, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lally RM, McNees P, Meneses K. Application of a novel transdisciplinary communication technique to develop an Internet-based psychoeducational program: CaringGuidance After Breast Cancer Diagnosis. Appl Nurs Res. 2015 Feb;28(1):e7-11. doi: 10.1016/j.apnr.2014.10.006. Epub 2014 Oct 31. PMID 25467063